CLINICAL TRIAL: NCT05624983
Title: Exploration of High Frequency Otoacoustic Emissions and Developmental Language Disorders
Acronym: OTOEMHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2022 SARRET
Record Dates: First submitted 2022-11-02; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-09

CONDITIONS: Language Development Disorders
Keywords: Language development disorders; otoemisions; child; high frequencies; hearing
MeSH Terms: conditions — Language Development Disorders | interventions — Otoscopy; Audiometry; Acoustic Impedance Tests

STUDY DESIGN:
Intervention Model Description: one group of cases (children with language disorder) one group of control (children without language disorder)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (children with language disorder) (Experimental): Hearing diagnostic test
  Interventions: Diagnostic Test: acoustic otoemisions; Diagnostic Test: Otoscopy; Diagnostic Test: Audiometry; Diagnostic Test: Tympanometry
- controle group (children without language disorder) (Other): Hearing diagnostic test
  Interventions: Diagnostic Test: acoustic otoemisions; Diagnostic Test: Otoscopy; Diagnostic Test: Audiometry; Diagnostic Test: Tympanometry

INTERVENTIONS:
Diagnostic Test: acoustic otoemisions — TOAE and DPOAE
Diagnostic Test: Otoscopy — presence of earwax checked by video otoscop
Diagnostic Test: Audiometry — Hearing Threshold will be measured with the AD528 interacoustics
Diagnostic Test: Tympanometry — Tympanic mobility will be measyred with the Titan interacoustics

SUMMARY:
Among the objective non-invasive audiological explorations the distorsion products of otoacoustic emissions (DPOAE) allow to quickly assess the function of the cochlear outer hair cells (without the active participation of the subject). This technique is used in newborn screening. While humans are able to perceive sounds in a frequency range of 20Hz to 20kHz, routine clinical audiological assessment is only concerned with frequencies between 1-4kHz.

This obscures the importance of high frequencies (HF) which can be easily assessed by DPOAEs. In young children, the perception of these high frequencies could also play an important role in language acquisition.

The main objective of this study is to evaluate the relationship between subtle high-frequency hearing impairment, as assessed by the DPOAE (non-invasive, rapid and simple audiological test), and language delay or difficulties in a pre-, peri- and school-age pediatric population.

ELIGIBILITY:
Inclusion Criteria for case (children with language disorder):

* Normal hearing (after an audiometry test, even if an ENT consultation has been carried out beforehand and if the doctor has not found any hearing problem, as defined in the NF EN ISO 70292017-04 standard, and according to an average hearing loss calculated according to the BIAP <20dB HL)
* Free and informed consent of the parental authority and the patient
* Affiliated to the social security system
* Presenting a developmental language acquisition disorder (score according to the EVALO / EVALEO test)
* For children between 15 and 17 years of age, completion of the EVALEO test before their 16th birthday

Inclusion Criteria for control (children without language disorder) :

* Normal hearing (after an audiometry test, even if an ENT consultation has been performed beforehand and if the doctor has not found any hearing problem, as defined in the NF EN ISO 70292017-04 standard, and according to an average hearing loss calculated according to the BIAP <20dB HL)
* Free and informed consent of the parental authority and the patient
* Enrolled in the social security system

Exclusion Criteria:

* Hearing disorder identified during the inclusion visit (presence of cerumen or foreign body in the earwax plug or foreign body in the external auditory canal, tympanometry suggesting a middle ear disorder, audiometry with thresholds outside the normal thresholds outside the normal range (0-20dB HL), absence of responses in (0-20dB HL), absence of responses in acoustic otoemissions or acoustic distortion products) on conversational frequencies between 500Hz and 4kHz.
* Declaration by the parents of an ENT follow-up for a hearing disorder and/or a speech therapy for a language disorder
* Refusal of participation evoked by the subject

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
HF DPOAE measurement | Day 1
  at frequencies 4265, 4688, 5154, 5666, 6229, 6847, 7527, 8275, 9096 and 10000 Hz

SECONDARY OUTCOMES:
Presence or absence of HF DPOAE | Day 1
  assessed by tympanometry, categorisation of this categorisation of this into 3 classes A, B and C frequency will be defined by a signal to noise ratio > 6 dB. The absence of DPOAE for each frequency will be defined by a signal to noise ratio ≤ 6 dB.
Functional status of the middle ear | Day 1
  assessed by tympanometry, categorisation of this categorisation of this into 3 classes A, B and C
Determination of the average hearing loss (baseline pure tone audiometry) | Day 1
  according to the BIAP, average of audiometric thresholds at 500Hz thresholds at 500Hz, 1kHz, 2kHz and 4kHz
Laterality of hearing loss at the DPOAE level with a classification into 3 groups | Day 1
  Not affected bilaterally affected, unilateral affected, bilateral affected; one side is considered to be affected if at least one of the at least one of the HF DPOAEs is ≤ 6 dB.
Severity and type of language impairment assessed by the EVALO/ EVALEO | day 1
  assessment and scoring by speech and language therapists

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, UMR INSERM 1107, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No